CLINICAL TRIAL: NCT01461785
Title: The Use of Activated Platelet Rich Plasma (PRP) in Human Autologous Fat Transfer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bergman Clinics (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, JCN Willemsen, MD, PhD candidate, Principal investigator of clinical research, Bergman Clinics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: JWJSLIPOFILLING
Record Dates: First submitted 2011-10-22; First posted 2011-10-28 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2012-07

CONDITIONS: Lipofilling; Human Autologous Fat Transfer
Keywords: Platelet rich plasma; Dermal improvement; Graft survival

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GROUP A: PRP + (Experimental): Group A (16 subjects) will receive lipofilling enriched with 3 ml of autologous PRP ( Platelet rich plasma) with lipofilling
  Interventions: Biological: Addition of PRP ( platelet rich plasma) to the lipograft; Procedure: Lipofilling of the midface
- GROUP B: PRP - (Placebo Comparator): Group B ( 16 subjects) will receive lipofilling without addition PRP. 27 ml blood will be drawn from the patient, but will be discarded, and not turned into PRP.
  Interventions: Procedure: Lipofilling of the midface

INTERVENTIONS:
Biological: Addition of PRP ( platelet rich plasma) to the lipograft — 27 ml blood will be drawn from the patient. The blood will be prepared according to the GPS System instructions (Biomet Biologics, LLC, Warsaw, Indiana USA). This desktop-size centrifuge has disposable cylinders to separate the different blood components (platelet rich plasma, PRP, platelet poor plasma, PPP, and red blood cells). The PRP is activated by adding calcium (15-volume % Ca2+ Sandoz®). creating activated Platelet Rich Plasma (aPRP).
  The lipograft of Group A will be enriched with 3ml of autologous PRP
  Arms: GROUP A: PRP +
Procedure: Lipofilling of the midface — The Coleman technique for fat harvesting and injection is employed but refined by utilizing a smaller, custom-made cannula for harvesting (inner diameter, 1.3 mm). The abdomen and upper legs are donor sites. Approximately two to three times more fat is harvested than the estimated amount required for the procedure. Fat is centrifuged for three minutes at the maximum speed of 3000 revolutions per minute after which the oil layer (top) and serum/infiltrate layer (bottom) are drained away, preserving the preadipocyte-rich pellet. Fat injection is performed in 1-mm aliquots with a short, curved Coleman cannula. Between 13 and 23 mL of fat is injected into the deep subcutaneous plane of each side of the face, except for the lower lid/tear trough region (where the injection is performed in the supraperiosteal/submuscular plane) and the temporal area (where the level of injection was above the superficial fascia of the temporal muscle).

SUMMARY:
In this prospective, randomized clinical trial, lipofilling of the midface with Platelet Rich Plasma (PRP) is compared with lipofilling of the midface without PRP. The main objective of this study is to investigate the effect of the addition of PRP to the autologous fat transfer on local skin quality improvement, graft survival, and recovery after the procedure.

DETAILED DESCRIPTION:
Soft tissue augmentation by the means of lipofilling is nowadays a frequently used technique in all forms of plastic surgery. In aesthetic facial surgery it has shown to increase the rejuvenating effect, in reconstructive surgery it has earned its place in the correction of soft tissue defects and athropy.

Post-operative loss of volume of the transplanted fat remains an uncertain factor in the procedure. In current literature, there are three main hypotheses on etiology of postoperative decrease in the graft volume; 1: the viability of the injected fat cells 2: impaired graft revascularization at the target site 3: the degree of fibrosis in the target area. Mentioned factors have limited the application of (large) volume lipotransfer.

Positive effects of lipofilling on skin quality have been reported. Coleman observed softening of wrinkles, decreasing pore size and pigmentation improvements on graft sites. Possible mechanisms of the claimed regenerative properties of the lipograft are explained by the high number of adipose derived stem cells. Although frequently described in literature, no objective results have been published to this date.

In this prospective study the investigators examine new methods in preventing postoperative volume loss by the addition of Platelet Rich Plasma (PRP), derived from the patients own blood, to the injected fat graft. The added PRP contains a wide range of growth factors for instance: Epidermal growth factor (EGF), Platelet derived growth factor (PDGF-AA), Transforming growth factor (TGF-B1, TGF-B2), Fibroblast growth factor (FGF) and Vascular endothelial growth factor (VEGF).

All previously mentioned factors have shown to play a key role in tissue regeneration after tissue damage. Especially VEGF is of great interest with the ability to promote neo-angiogenesis in the graft, and thus, in theory, reducing fat necrosis and seroma formation.

Current, scientifically validated, use of PRP include treatment of chronic and soft tissue ulcerations, applications in the periodontal and oral surgery, maxillofacial surgery, orthopaedic and trauma surgery, cosmetic and plastic surgery, spinal surgery, heart bypass surgery, and burns. In all mentioned applications, PRP showed to have a positive influence on the tissue recovery and regeneration. Local PRP application in damaged animal and human skin showed to have regenerative properties. Structural changes to the dermal layer were observed in biopsies.

In this prospective, randomized clinical trial, lipofilling of the midface with PRP is compared with lipofilling of the midface without PRP. The main objective of this study is to investigate the effect of the addition of PRP to the autologous fat transfer on local skin quality improvement, graft survival, and recovery after the procedure.

The synergy achieved by lipofilling with PRP may hold many future applications in both reconstructive and aesthetic plastic surgery. Current limitation of lipofilling, especially large volume lipo transfer (allowing reconstruction in one procedure in stead of multiple with smaller volumes) and lipofilling in pour vascularised tissue (eg. fibrosis after radiation therapy) may be countered by the addition of PRP. Furthermore, the suggested local skin improvements could be used in scar revisions and burn treatment in the future, bypassing invasive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged 30-65
* Stable normal BMI (20-25) (1 year stable between 20-25)

Exclusion Criteria:

•• Male

* Aged below 30 or above 65 years
* Aged between 45 and 55 and in the menopause
* Aged between 55 and 65 and pre-menopause
* Prior operations in the mid-face
* Any oncological event in the patients history
* A known psychiatric condition
* A known systemic disease that will impair wound healing ( eg diabetus mellitus, known atherosclerosis with an event that required hospitalization, collagen diseases, diseases of the skin).
* Smoking
* 20<BMI<25 or an unstable BMI: 1 year plus-minus 5 points.
* Pregnancy or active child wish
* Frequent exposure to known carcinogenic substances ( eg. work related).
* Active or previous use of hormone replacement therapy.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Cutometry | 1 year post-operative of the last included patient, estimate is 18 months
  Postoperative skin quality measured with a Multi Probe Adapter system (Courage Khanza Colone Germany) containing several skin measurement probes (Maxameter mx18: Assessing melanin content and erythema level, Tewameter TM300: Skin barrier function and transepidermal waterloss, Cutometer MPA580: Mechanical parameters of the skin) on predetermined fixed positions in the face on predetermined times . (pre-operative, 1 week postoperative, 3 months post-operative and 1 year post-operative.)

SECONDARY OUTCOMES:
Panel assessment | 1 year post-operative of the last included patient, estimate is 18 months
  Standardized photos will be taken pre-, and post-operatively ( at 3 months and 1 year follow-up ) The photos will be analysed by two separate panels using validated scoring systems ( an adapted Moolenburg and Strasser). Both questionnaires will focus on changes in facial volume. The panels will consist of five independent plastic surgeons and five laypersons (all blinded).(pre-operative, 3 months post-operative and 1 year post-operative.)
Patient questionnaire | 1 year post-operative of the last included patient, estimate is 18 months
  Analysis of a patient questionnaire sent at 4 weeks post-operative, with number of complications, recovery time (return to work/ return to social activity) and patient self-assessment (visual analogue score) as main endpoints. This questionnaire will use the standardized FACE-Q list that will be published in the fourth quarter of 2011. Use of topical skin products and sun exposure will be added to this questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Stevens, MD, PhD, Study Director — Bergman Clinics; Joep Willemsen, MD, Principal Investigator — Bergman Clinics
Locations (1):
- Bergman Clinics, The Hague, South Holland, Netherlands

REFERENCES:
- [Background] Little JW. Applications of the classic dermal fat graft in primary and secondary facial rejuvenation. Plast Reconstr Surg. 2002 Feb;109(2):788-804. doi: 10.1097/00006534-200202000-00059. PMID 11818872
- [Background] Coleman SR. Facial recontouring with lipostructure. Clin Plast Surg. 1997 Apr;24(2):347-67. PMID 9142473
- [Background] Tzikas TL. Lipografting: autologous fat grafting for total facial rejuvenation. Facial Plast Surg. 2004 May;20(2):135-43. doi: 10.1055/s-2004-861754. PMID 15643580
- [Background] Clauser L, Polito J, Mandrioli S, Tieghi R, Denes SA, Galie M. Structural fat grafting in complex reconstructive surgery. J Craniofac Surg. 2008 Jan;19(1):187-91. doi: 10.1097/scs.0b013e31815c94f5. PMID 18216687
- [Background] Ducic Y, Pontius AT, Smith JE. Lipotransfer as an adjunct in head and neck reconstruction. Laryngoscope. 2003 Sep;113(9):1600-4. doi: 10.1097/00005537-200309000-00036. PMID 12972941
- [Background] Jackson IT, Simman R, Tholen R, DiNick VD. A successful long-term method of fat grafting: recontouring of a large subcutaneous postradiation thigh defect with autologous fat transplantation. Aesthetic Plast Surg. 2001 May-Jun;25(3):165-9. doi: 10.1007/s002660010115. PMID 11426305
- [Background] Conde-Green A, Baptista LS, de Amorin NF, de Oliveira ED, da Silva KR, Pedrosa Cda S, Borojevic R, Pitanguy I. Effects of centrifugation on cell composition and viability of aspirated adipose tissue processed for transplantation. Aesthet Surg J. 2010 Mar;30(2):249-55. doi: 10.1177/1090820X10369512. PMID 20442104
- [Background] Erdim M, Tezel E, Numanoglu A, Sav A. The effects of the size of liposuction cannula on adipocyte survival and the optimum temperature for fat graft storage: an experimental study. J Plast Reconstr Aesthet Surg. 2009 Sep;62(9):1210-4. doi: 10.1016/j.bjps.2008.03.016. Epub 2008 Jun 20. PMID 18572007
- [Background] Nguyen A, Pasyk KA, Bouvier TN, Hassett CA, Argenta LC. Comparative study of survival of autologous adipose tissue taken and transplanted by different techniques. Plast Reconstr Surg. 1990 Mar;85(3):378-86; discussion 387-9. PMID 2304989
- [Background] Nishimura T, Hashimoto H, Nakanishi I, Furukawa M. Microvascular angiogenesis and apoptosis in the survival of free fat grafts. Laryngoscope. 2000 Aug;110(8):1333-8. doi: 10.1097/00005537-200008000-00021. PMID 10942136
- [Background] Yamaguchi M, Matsumoto F, Bujo H, Shibasaki M, Takahashi K, Yoshimoto S, Ichinose M, Saito Y. Revascularization determines volume retention and gene expression by fat grafts in mice. Exp Biol Med (Maywood). 2005 Nov;230(10):742-8. doi: 10.1177/153537020523001007. PMID 16246901
- [Background] Sommer B, Sattler G. Current concepts of fat graft survival: histology of aspirated adipose tissue and review of the literature. Dermatol Surg. 2000 Dec;26(12):1159-66. PMID 11134994
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Nikolidakis D, Jansen JA. The biology of platelet-rich plasma and its application in oral surgery: literature review. Tissue Eng Part B Rev. 2008 Sep;14(3):249-58. doi: 10.1089/ten.teb.2008.0062. PMID 18601587
- [Background] Eppley BL, Pietrzak WS, Blanton M. Platelet-rich plasma: a review of biology and applications in plastic surgery. Plast Reconstr Surg. 2006 Nov;118(6):147e-159e. doi: 10.1097/01.prs.0000239606.92676.cf. PMID 17051095
- [Background] Ferrara N, Gerber HP. The role of vascular endothelial growth factor in angiogenesis. Acta Haematol. 2001;106(4):148-56. doi: 10.1159/000046610. PMID 11815711
- [Background] Nakamura S, Ishihara M, Takikawa M, Murakami K, Kishimoto S, Nakamura S, Yanagibayashi S, Kubo S, Yamamoto N, Kiyosawa T. Platelet-rich plasma (PRP) promotes survival of fat-grafts in rats. Ann Plast Surg. 2010 Jul;65(1):101-6. doi: 10.1097/SAP.0b013e3181b0273c. PMID 20548232
- [Background] Ono S, Ogawa R, Hyakusoku H. Re: Use of Aquamid as a filler for facial rejuvenation in orientals. J Plast Reconstr Aesthet Surg 2009;62:1245-9. J Plast Reconstr Aesthet Surg. 2010 Jul;63(7):1227-8. doi: 10.1016/j.bjps.2009.12.008. Epub 2010 Jan 12. No abstract available. PMID 20061200
- [Background] Salemi S, Rinaldi C, Manna F, Guarneri GF, Parodi PC. Reconstruction of lower leg skin ulcer with autologous adipose tissue and platelet-rich plasma. J Plast Reconstr Aesthet Surg. 2008 Dec;61(12):1565-7. doi: 10.1016/j.bjps.2008.04.048. Epub 2008 Aug 10. No abstract available. PMID 18694662
- [Background] Lindeboom JA, Mathura KR, Aartman IH, Kroon FH, Milstein DM, Ince C. Influence of the application of platelet-enriched plasma in oral mucosal wound healing. Clin Oral Implants Res. 2007 Feb;18(1):133-9. doi: 10.1111/j.1600-0501.2006.01288.x. PMID 17224034
- [Background] Shashikiran ND, Reddy VV, Yavagal CM, Zakirulla M. Applications of platelet-rich plasma (PRP) in contemporary pediatric dentistry. J Clin Pediatr Dent. 2006 Summer;30(4):283-6. doi: 10.17796/jcpd.30.4.8663xu2610324v36. PMID 16937851
- [Background] Pietrzak WS, Eppley BL. Platelet rich plasma: biology and new technology. J Craniofac Surg. 2005 Nov;16(6):1043-54. doi: 10.1097/01.scs.0000186454.07097.bf. PMID 16327552
- [Background] El-Sharkawy H, Kantarci A, Deady J, Hasturk H, Liu H, Alshahat M, Van Dyke TE. Platelet-rich plasma: growth factors and pro- and anti-inflammatory properties. J Periodontol. 2007 Apr;78(4):661-9. doi: 10.1902/jop.2007.060302. PMID 17397313
- [Background] Wrotniak M, Bielecki T, Gazdzik TS. Current opinion about using the platelet-rich gel in orthopaedics and trauma surgery. Ortop Traumatol Rehabil. 2007 May-Jun;9(3):227-38. English, Polish. PMID 17721419
- [Background] Mishra A, Woodall J Jr, Vieira A. Treatment of tendon and muscle using platelet-rich plasma. Clin Sports Med. 2009 Jan;28(1):113-25. doi: 10.1016/j.csm.2008.08.007. PMID 19064169
- [Background] Bhanot S, Alex JC. Current applications of platelet gels in facial plastic surgery. Facial Plast Surg. 2002 Feb;18(1):27-33. doi: 10.1055/s-2002-19824. PMID 11823930
- [Background] Henderson JL, Cupp CL, Ross EV, Shick PC, Keefe MA, Wester DC, Hannon T, McConnell D. The effects of autologous platelet gel on wound healing. Ear Nose Throat J. 2003 Aug;82(8):598-602. PMID 14503096
- [Background] Redaelli A, Romano D, Marciano A. Face and neck revitalization with platelet-rich plasma (PRP): clinical outcome in a series of 23 consecutively treated patients. J Drugs Dermatol. 2010 May;9(5):466-72. PMID 20480789
- [Background] Engebretsen L, Steffen K, Alsousou J, Anitua E, Bachl N, Devilee R, Everts P, Hamilton B, Huard J, Jenoure P, Kelberine F, Kon E, Maffulli N, Matheson G, Mei-Dan O, Menetrey J, Philippon M, Randelli P, Schamasch P, Schwellnus M, Vernec A, Verrall G. IOC consensus paper on the use of platelet-rich plasma in sports medicine. Br J Sports Med. 2010 Dec;44(15):1072-81. doi: 10.1136/bjsm.2010.079822. No abstract available. PMID 21106774
- [Background] Wang-Saegusa A, Cugat R, Ares O, Seijas R, Cusco X, Garcia-Balletbo M. Infiltration of plasma rich in growth factors for osteoarthritis of the knee short-term effects on function and quality of life. Arch Orthop Trauma Surg. 2011 Mar;131(3):311-7. doi: 10.1007/s00402-010-1167-3. Epub 2010 Aug 17. PMID 20714903
- [Background] Donofrio LM. Panfacial volume restoration with fat. Dermatol Surg. 2005 Nov;31(11 Pt 2):1496-505. doi: 10.2310/6350.2005.31234. PMID 16416631
- [Background] Eremia S, Newman N. Long-term follow-up after autologous fat grafting: analysis of results from 116 patients followed at least 12 months after receiving the last of a minimum of two treatments. Dermatol Surg. 2000 Dec;26(12):1150-8. PMID 11134993
- [Background] Ersek RA. Transplantation of purified autologous fat: a 3-year follow-up is disappointing. Plast Reconstr Surg. 1991 Feb;87(2):219-27; discussion 228. PMID 1750860
- [Background] Brucker M, Sati S, Spangenberger A, Weinzweig J. Long-term fate of transplanted autologous fat in a novel rabbit facial model. Plast Reconstr Surg. 2008 Sep;122(3):749-754. doi: 10.1097/PRS.0b013e3181815a41. PMID 18766037
- [Background] Lacci KM, Dardik A. Platelet-rich plasma: support for its use in wound healing. Yale J Biol Med. 2010 Mar;83(1):1-9. PMID 20351977
- [Background] Tischler M. Platelet rich plasma. The use of autologous growth factors to enhance bone and soft tissue grafts. N Y State Dent J. 2002 Mar;68(3):22-4. PMID 11989332
- [Background] Strem BM, Hicok KC, Zhu M, Wulur I, Alfonso Z, Schreiber RE, Fraser JK, Hedrick MH. Multipotential differentiation of adipose tissue-derived stem cells. Keio J Med. 2005 Sep;54(3):132-41. doi: 10.2302/kjm.54.132. PMID 16237275
- [Background] Gimble J, Guilak F. Adipose-derived adult stem cells: isolation, characterization, and differentiation potential. Cytotherapy. 2003;5(5):362-9. doi: 10.1080/14653240310003026. PMID 14578098
- [Background] Madonna R, Geng YJ, De Caterina R. Adipose tissue-derived stem cells: characterization and potential for cardiovascular repair. Arterioscler Thromb Vasc Biol. 2009 Nov;29(11):1723-9. doi: 10.1161/ATVBAHA.109.187179. Epub 2009 Jul 23. PMID 19628786
- [Background] Kim JH, Jung M, Kim HS, Kim YM, Choi EH. Adipose-derived stem cells as a new therapeutic modality for ageing skin. Exp Dermatol. 2011 May;20(5):383-7. doi: 10.1111/j.1600-0625.2010.01221.x. Epub 2011 Feb 28. PMID 21355887
- [Background] Pallua N, Wolter T, Markowicz M. Platelet-rich plasma in burns. Burns. 2010 Feb;36(1):4-8. doi: 10.1016/j.burns.2009.05.002. Epub 2009 Jun 21. PMID 19541423
- [Background] Strasser EJ. Application of an objective grading system for the evaluation of cosmetic surgical results. Plast Reconstr Surg. 2002 Apr 15;109(5):1733-40. doi: 10.1097/00006534-200204150-00042. No abstract available. PMID 11932628
- [Background] Pusic AL, Klassen AF, Scott AM, Cano SJ. Discussion. The measure of face-lift patient satisfaction: the Owsley Facelift Satisfaction Survey with a long-term follow-up study. Plast Reconstr Surg. 2010 Jul;126(1):258-260. doi: 10.1097/PRS.0b013e3181dbba19. No abstract available. PMID 20595872
- [Background] Nedelec B, Correa JA, Rachelska G, Armour A, LaSalle L. Quantitative measurement of hypertrophic scar: interrater reliability and concurrent validity. J Burn Care Res. 2008 May-Jun;29(3):501-11. doi: 10.1097/BCR.0b013e3181710881. PMID 18388576
- [Background] Draaijers LJ, Botman YA, Tempelman FR, Kreis RW, Middelkoop E, van Zuijlen PP. Skin elasticity meter or subjective evaluation in scars: a reliability assessment. Burns. 2004 Mar;30(2):109-14. doi: 10.1016/j.burns.2003.09.003. PMID 15019116
- [Background] Ryu HS, Joo YH, Kim SO, Park KC, Youn SW. Influence of age and regional differences on skin elasticity as measured by the Cutometer. Skin Res Technol. 2008 Aug;14(3):354-8. doi: 10.1111/j.1600-0846.2008.00302.x. PMID 19159383
- [Background] Ezure T, Hosoi J, Amano S, Tsuchiya T. Sagging of the cheek is related to skin elasticity, fat mass and mimetic muscle function. Skin Res Technol. 2009 Aug;15(3):299-305. doi: 10.1111/j.1600-0846.2009.00364.x. PMID 19624426
- [Background] Tronnier H, Wiebusch M, Heinrich U. Change in skin physiological parameters in space--report on and results of the first study on man. Skin Pharmacol Physiol. 2008;21(5):283-92. doi: 10.1159/000148045. Epub 2008 Jul 28. PMID 18663342
- [Background] Yamaguchi R, Terashima H, Yoneyama S, Tadano S, Ohkohchi N. Effects of platelet-rich plasma on intestinal anastomotic healing in rats: PRP concentration is a key factor. J Surg Res. 2012 Apr;173(2):258-66. doi: 10.1016/j.jss.2010.10.001. Epub 2010 Nov 2. PMID 21074782
- [Background] Krupski WC, Reilly LM, Perez S, Moss KM, Crombleholme PA, Rapp JH. A prospective randomized trial of autologous platelet-derived wound healing factors for treatment of chronic nonhealing wounds: a preliminary report. J Vasc Surg. 1991 Oct;14(4):526-32; discussion 532-6. PMID 1920650
- [Background] Silva A, Sampaio R. Anatomic ACL reconstruction: does the platelet-rich plasma accelerate tendon healing? Knee Surg Sports Traumatol Arthrosc. 2009 Jun;17(6):676-82. doi: 10.1007/s00167-009-0762-8. Epub 2009 Mar 14. PMID 19288080
- [Background] de Jonge S, de Vos RJ, Van Schie HT, Verhaar JA, Weir A, Tol JL. One-year follow-up of a randomised controlled trial on added splinting to eccentric exercises in chronic midportion Achilles tendinopathy. Br J Sports Med. 2010 Jul;44(9):673-7. doi: 10.1136/bjsm.2008.052142. Epub 2008 Oct 6. PMID 18838406
- [Background] Dogramaci Y, Kalaci A, Savas N, Duman IG, Yanat AN. Treatment of lateral epicondilitis using three different local injection modalities: a randomized prospective clinical trial. Arch Orthop Trauma Surg. 2009 Oct;129(10):1409-14. doi: 10.1007/s00402-009-0832-x. Epub 2009 Feb 14. PMID 19219442
- [Background] Peerbooms JC, Sluimer J, Bruijn DJ, Gosens T. Positive effect of an autologous platelet concentrate in lateral epicondylitis in a double-blind randomized controlled trial: platelet-rich plasma versus corticosteroid injection with a 1-year follow-up. Am J Sports Med. 2010 Feb;38(2):255-62. doi: 10.1177/0363546509355445. PMID 20448192
- [Background] Martinez-Zapata MJ, Marti-Carvajal A, Sola I, Bolibar I, Angel Exposito J, Rodriguez L, Garcia J. Efficacy and safety of the use of autologous plasma rich in platelets for tissue regeneration: a systematic review. Transfusion. 2009 Jan;49(1):44-56. doi: 10.1111/j.1537-2995.2008.01945.x. Epub 2008 Oct 14. PMID 18954394